CLINICAL TRIAL: NCT06281574
Title: What Are the Determinants for Return to Work After Shoulder Arthroplasty
Brief Title: What Are the Determinants for RTW After SA
Acronym: RTW after SA
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S67346
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Arthroplasty
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with shoulder arthroplasty: Including all surgical interventions (anatomic total shoulder arthroplasty, humeral head hemi arthroplasty or reversed shoulder arthroplasty) for patients with shoulder arthroplasty
  Interventions: Procedure: Questionnaires

INTERVENTIONS:
Procedure: Questionnaires — To assess the shoulder function, the following questionnaires will be used:
  The validated Dutch translation of the Oxford Shoulder Score (OSS) The validated Dutch translation of the Simple Shoulder Test (SST) The Subjective Shoulder Value (SVV) To assess the work ability patients will use the validated Dutch work-related questionnaire for upper extremity disorders (WORQ-UP)

SUMMARY:
Shoulder arthroplasty is becoming increasingly common, due to ageing of the population. Historically, surgeons have been reluctant to use a shoulder replacement in younger patients. During the last decades however, there was an improvement of surgical techniques and implants which resulted in the fact that these procedures are nowadays more frequently used in younger patients. Combined with the increasing life expectancy and the increased age of retirement, both elderly and younger patients hope to continue their jobs after prosthetic replacement.

Recent literature shows that the majority patients is able to resume their work following shoulder arthroplasty.

This study aims to analyze the RTW percentage in a Belgian cohort of patients with a shoulder replacement. This study hopes to identify factors that might influence the RTW.

DETAILED DESCRIPTION:
Shoulder arthroplasty is becoming increasingly common, due to ageing of the population. Historically, surgeons have been reluctant to use a shoulder replacement in younger patients, due to the high incidence of complications and the limited longevity of the implant. Therefore, this type of surgery remained reserved for the elderly patients. During the last decades however, improvement of surgical techniques and implants have made it possible to expand the indications for anatomical total shoulder arthroplasty (aTSA), humeral head hemi-arthroplasty (HHA) and reversed total shoulder arthroplasty (rTSA), resulting in significant improvements in range of motion, functional outcomes, quality of life and reported pain scores. As a result, these procedures are nowadays more frequently used in younger patients. Combined with the increasing life expectancy and the increased age of retirement, both elderly and younger patients hope to continue their jobs after prosthetic replacement.

Recent literature shows that the majority patients is able to resume their work following shoulder arthroplasty.

This study aims to analyze the RTW percentage in a Belgian cohort of patients with a shoulder replacement. This study hopes to identify factors that might influence the RTW. An enhanced understanding of this social, medical and economic issue will enable surgeons to give more tailored advice to their patients regarding RTW after shoulder replacement surgery and accordingly reduce the economic burden on Belgian society.

ELIGIBILITY:
Inclusion Criteria:

* Current evidence suggests that no significant changes in functionality can be expected 2 years after surgery. Therefore, we will include patients who were operated between January 2010 and January 2022 at the University Hospital Leuven
* Patients ≥ 18 years old and ≤ 63 years old at time of surgery
* Implantation of an anatomic total shoulder arthroplasty, humeral head hemi arthroplasty or reversed shoulder arthroplasty

Exclusion Criteria:

* Age < 18 and > 63 years at time of surgery
* Limited knowledge of Dutch

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Population of patients with a shoulder arthroplasty surgery between January 2010 and January 2022 at University Hospitals Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Return to work | Baseline
  Collection how many of the study participants will return to work after a shoulder arthroplasty. This question is answered with yes or no.

SECONDARY OUTCOMES:
Type of shoulder arthroplasty | Baseline
  Collect how many participants received an anatomic total shoulder arthroplasty (aTSA), reverse total shoulder arthroplasty (rTSA) or humeral hemi-arthroplasty (HHA)
WORQ-UP (work-related questionnaire for upper extremity disorders) | Baseline
  A questionnaire used to identify self-reported difficulty performing common work-related tasks. It consists of 17 items.
SSV (Subjective Shoulder Value) | Baseline
  Question to subjectively evaluate a patient's shoulder function. Which percentage do you give your shoulder. A normal shoulder is 100% and worst schoulder is 0%.
SST (Dutch translation of the Simple Shoulder Test) | Baseline
  A questionnaire that contains 12 items to be answered by the patient independently: 2 about function related to pain, 7 about function/strength, and 3 about range of motion. Questions are answered by yes or no. A final score of 0 = worst and 12 = best. Scores are subsequently transformed by number of 'yes' items/ number of completed items x 100 = % 'yes' responses. A final score of 0= worst function and 100= best function.
OSS (Oxford Shoulder Score) | Baseline
  A questionnaire that contains 12 items to be answered by the patient independently. There are 5 categories of response for every question, corresponding to a score ranging from 1 to 5. Scores are combined to give a single score, with a range from 12 (best) to 60 (worst). The questions deal with pain (degree, time point) and possible handicaps in private and professional life. It is divided 20/40 corresponding to pain/activities of daily living.
Self-made questionnaire | Baseline
  A questionnaire where the participants is asked if they returned back to their jobs and if so how many months after surgery, what their job satisfaction is, if work-related adaptations were made by the employer to ease the return to work process, what their marital status and educational qualifications are.
Belgisch Kenniscentrum over welzijn op het werk (BeSWIC) | Baseline
  The participants' occupations is classified as light, medium, hard or very hard occupation

CONTACTS AND LOCATIONS:
Overall Officials: Filip Verhaegen, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No